CLINICAL TRIAL: NCT03570359
Title: A Randomised, Double-blind, Placebo-controlled Study, in COPD Patients With and Without a Confirmed Respiratory Virus Infection Assessing Anti-viral Biomarker Responses and Clinical Effects of Inhaled SNG001 Compared to Placebo
Brief Title: A Study to Test a Potential New Treatment for COPD Patients Suffering From the Common Cold or Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synairgen Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG015; 2017-003679-75 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-06-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will be randomised to one of two treatment groups (SNG001 or placebo).
  In Part 1 the ratio will be 4:1 and in Part 2 the ratio will be 1:1, both according to a pre-specified randomisation schedule. In Part 2, prior to randomisation to SNG001 or placebo, patients will be stratified into two groups; those with cold symptoms without a moderate COPD exacerbation (Group A), and those who have a moderate COPD exacerbation with or without cold symptoms (Group B).
  For both parts of the study, patients will be randomised according to a pre-specified randomisation schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon beta 1a (Active Comparator): Part 1- Interferon beta 1a once a day for 3 days via inhalation
  Part 2 - Interferon beta 1a once a day for 14 days via inhalation
  Interventions: Drug: Interferon Beta-1A
- Placebo (Placebo Comparator): Part 1- placebo once a day for 3 days via inhalation
  Part 2 - placebo once a day for 14 days via inhalation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Interferon Beta-1A — Interferon Beta-1A via inhalation
  Other Names: SNG001
  Arms: Interferon beta 1a
Other: Placebo — Placebo via inhalation
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the safety of inhaled SNG001 and the ability of inhaled SNG001 to 'switch on' the cells' anti-viral defences in patients with chronic obstructive pulmonary disease (COPD). The study consist of two parts.

Part 1 will assess the safety of inhaled SNG001 in ten patients with stable COPD.

Part 2 will assess efficacy and safety of inhaled SNG001 in 120 patients with COPD with a cold or COPD exacerbation.

DETAILED DESCRIPTION:
When people with COPD get a respiratory virus such as a cold or flu it often increases their COPD symptoms, leading them to require treatment with either antibiotics or oral steroids and severely affecting their quality of life. SNG001 is the study medication, and it contains interferon beta (interferon-β) which is a natural antiviral protein. In this study we will look to see whether inhaled SNG001 can boost anti-viral responses and minimise the worsening of COPD symptoms/lung function when patients have a confirmed respiratory virus.

In Part 1 ten COPD patients without a respiratory virus will be randomised to receive three days of SNG001 or placebo. The aim of this part of the study is to assess safety of SNG001 in COPD patients.

In Part 2 COPD patients will contact the research team when they experience cold or flu symptoms or a deterioration of their COPD symptoms. At this point, eligible patients will undergo a virus detection test and those that test positive for a virus will be randomised 1:1 to receive SNG001 or placebo once daily for 14 days. The first dose of study medication will be administered within 48 hours. Other assessments will be performed during the 14 days of treatment to look for changes in anti-viral biomarkers, lung function and COPD symptoms. Patients will also be followed up 14 days post end of treatment.

ELIGIBILITY:
PART 1 - Inclusion Criteria:

1. Male or female, between and including 40-75 years of age, at the time of the screening visit.
2. A confirmed physician diagnosis of COPD or a medical history consistent with a diagnosis of COPD for at least 12 months prior to the screening visit.
3. Post-bronchodilator FEV1 ≥40% of predicted and FEV1/FVC ratio <0.7 (at screening).
4. FEV1 ≥30% of predicted (at Visit 2, pre-dose).
5. Should have stable COPD, having no symptoms of an exacerbation and/or respiratory tract infection currently and/or within the past 6 weeks of screening and/or randomisation.
6. Should be prescribed and taking regularly one or more long acting bronchodilators (e.g. long acting β2 agonist [LABA], long acting muscarinic antagonist [LAMA]) with or without an inhaled corticosteroid maintenance therapy for their COPD.
7. Patients who produce sputum most days.
8. Provide written informed consent.
9. The patient produced an adequate sputum sample at the screening visit.
10. Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception. Women should have been stable on their chosen method of birth control for a minimum of 3 months before entering the trial and should continue with birth control for 1 month after the last dose. In addition to the acceptable birth control method (except for the practice of total sexual abstinence), condom (in UK with spermicides) should be used by the male partner for sexual intercourse from randomisation (Visit 2) and for 1 month after the last dose to prevent pregnancy.

    Women of childbearing potential must have a negative pregnancy test at screening and prior to randomisation.

    Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomisation without an alternative medical cause. The following age specific requirements apply:
    * Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and if follicle stimulating hormone (FSH) levels are in the postmenopausal range. If the FSH result is not available at the time of randomization, the patient must have a negative pregnancy test and agree to use highly effective contraception methods until the FSH result is available.
    * Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
11. Motivation (in the Investigator's opinion) to comply with protocol requirements and complete all study visits, including the ability to communicate well with the Investigator and be capable of understanding the nature of the research and its treatment (including its risks and potential benefits).

PART 2 - pre-treatment Inclusion Criteria:

1. Male or female, between and including 40-85 years of age at the time of the consent visit.
2. A confirmed physician diagnosis of COPD or a medical history consistent with a diagnosis of COPD for at least 12 months prior to the consent visit.
3. Current or ex-smoker with ≥ 10 pack years of smoking history.
4. Post bronchodilator FEV1/FVC ratio <0.7.
5. Post bronchodilator FEV1 ≥40% of the predicted value. Once the safety data for the first 16 patients have been reviewed and approved by the DSMC the criterion will be changed to a post bronchodilator of FEV1 ≥30% of the predicted value*.
6. To have had 1 or more COPD exacerbations in the last 12 months requiring intervention with oral corticosteroids and/or antibiotics.
7. Patient reported evidence that a respiratory virus has made their COPD significantly worse in the past.
8. Should be prescribed and taking regularly one or more long acting bronchodilator (e.g. long acting β2 agonist [LABA], long acting muscarinic antagonist [LAMA]) with or without an inhaled corticosteroid maintenance therapy for their COPD.
9. Patients on self-management plans agree to consult a healthcare professional prior to taking oral corticosteroids or antibiotics for treatment of a COPD exacerbation.
10. Provide written informed consent.
11. Be the owner of a mobile phone, and be able to, and agree to, respond to the required SMS (text) messages for the trial.
12. Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception. Acceptable birth control methods are tubal occlusion, intrauterine device (provided coils are copper-banded), levonorgestrel intrauterine system (eg, Mirena™), medroxyprogesterone injections (eg, Depo- Provera™), etonogestrel implants (eg, Implanon™, Norplan™), normal and low dose combined oral pills, norelgestromin / ethinylestradiol transdermal system, intravaginal device (eg, ethinylestradiol and etonogestrel ), desogestrel (eg, Cerazette™), total sexual abstinence and vasectomised sexual partner. Women should have been stable on their chosen method of birth control for a minimum of 3 months before entering the trial and should continue with birth control for 1 month after the last dose of inhaled IFN-β-1a/matching placebo. In addition to the acceptable birth control method (except for the practice of total sexual abstinence), condom (in UK with spermicides) should be used by the male partner for sexual intercourse from randomisation (Visit 2) and for 1 month after the last dose of inhaled IFN-β-1a/matching placebo to prevent pregnancy.

    Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomisation without an alternative medical cause. The following age specific requirements apply:
    * Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and if FSH levels are in the postmenopausal range.
    * Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
13. Motivation (in the Investigator's opinion) to comply with protocol requirements and complete all study visits, including the ability to communicate well with the Investigator and be capable of understanding the nature of the research and its treatment (including its risks and potential benefits).

    * patients will continue to be recruited using the inclusion criterion FEV1 ≥40%, until the change to FEV1 ≥30% has been approved by the DSMC.

PART 1 - Exclusion Criteria:

1. Any condition, including findings in the medical history or in the pre-randomisation assessments that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the patient in the study or that could interfere with the study objectives, conduct or evaluation.
2. Current treatment or treatment within the past 6 weeks with oral corticosteroids.
3. Oxygen saturation of ≤ 92%.
4. Patients who require any form of oxygen therapy or non-invasive ventilation.
5. The patient has received live/attenuated vaccines in the past six weeks prior to randomisation or inactivated/killed, subunit or conjugate vaccines in the past two weeks prior to randomisation.
6. Current or previous participation in another clinical trial where the patient has received a dose of an investigational medicinal product (IMP) containing small molecules within 12 weeks prior to entry into this study or containing biologicals within 12 months prior to entry into this study.
7. Active interstitial lung disease or past history of lung cancer not considered cured, significant bronchiectasis, cystic fibrosis, alpha-1 antitrypsin deficiency or a history of significant chronic asthma.
8. Patients who currently have, or have had within the past 3 months, any significant underlying medical condition(s) that could impact the interpretation of results (e.g. non respiratory infections, haematological disease, malignancy, renal disease, hepatic disease, coronary heart disease or other cardiovascular disease [including arrhythmias], endocrine or gastrointestinal disease).
9. History of hypersensitivity to natural or recombinant IFN-β or to any of the excipients in the drug preparation.
10. Significant history of depressive disorder or suicidal ideation. Specifically, individuals with current severe depression (i.e. a low mood, which pervades all aspects of life and an inability to experience pleasure in activities that formerly were enjoyed); individuals with a past history of depression that required hospitalisation or referral to psychiatric services in the past 5 years; individuals who currently feel suicidal or have attempted suicide in the past.
11. Patients who are currently receiving anti-epileptic therapy and/or have uncontrolled epilepsy.
12. History of drug or alcohol abuse within 12 months prior to enrolment.
13. Female who is breast-feeding, pregnant or intends to become pregnant.
14. Patients with clinically significant arrhythmias or implantation of permanent pacemaker or implanted cardiac defibrillator.
15. Patients with unstable ischaemic heart disease (including, but not limited to, unstable angina or myocardial infarction) or stroke within the preceding 6 months.

PART 2 - Pre-treatment Exclusion Criteria:

1. Any condition, including findings in the medical history or in the pre-study assessments, or any treatment, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the patient in the study or that could interfere with the study objectives, conduct or evaluation.
2. The patient currently has a moderate or severe exacerbation of COPD.
3. The patient had a moderate or severe exacerbation of COPD that resolved less than 2 weeks ago (with resolution defined as return to patient's baseline COPD symptoms or the Investigator does not expect any further improvement of patient's symptoms).
4. The patient stopped taking treatment (antibiotics and/or oral corticosteroids) for an exacerbation of COPD less than 2 weeks ago.
5. The patient currently has an upper or lower respiratory tract infection.
6. Oxygen saturation of ≤92% .
7. Patients who require long-term oxygen therapy.
8. Current or previous participation in another clinical trial where the patient has received a dose of an IMP containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study.
9. Active interstitial lung disease or past history of lung cancer not considered cured, significant bronchiectasis, cystic fibrosis, alpha-1 antitrypsin deficiency or a history of significant chronic asthma.
10. Patients who currently have, or have had within the past 3 months, any significant underlying medical condition(s) that could impact interpretation of results (e.g. non respiratory infections, haematological disease, malignancy, renal disease, hepatic disease, coronary heart disease or other cardiovascular disease [including arrhythmias], endocrine or gastrointestinal disease).
11. History of hypersensitivity to natural or recombinant IFN-β or to any of the excipients in the drug preparation.
12. Significant history of depressive disorder or suicidal ideation. Specifically, individuals with current severe depression (i.e. a low mood, which pervades all aspects of life and an inability to experience pleasure in activities that formerly were enjoyed); individuals with a past history of depression that required hospitalisation or referral to psychiatric services in the past 5 years; individuals who currently feel suicidal or have attempted suicide in the past 5 years.
13. Patients who are currently receiving anti-epileptic therapy and/or have uncontrolled epilepsy.
14. History of drug or alcohol abuse within 12 months prior to enrolment .
15. Female who is breast-feeding, lactating, pregnant or intends to become pregnant.
16. Patients with clinically significant arrhythmias or implantation of permanent pacemaker or implanted cardiac defibrillator.
17. Patients with unstable ischaemic heart disease (including, but not limited to, unstable angina or myocardial infarction) or stroke within the preceding 6 months.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | from Baseline (pre-treatment on day 1) to day 3
  Part 1
Peak Expiratory Flow Rate (PEFR) | from Baseline (pre-treatment on day 1) to day 3
  Part 1
Anti-viral IFN-stimulated genes in cells from expectorated sputum. | from Baseline (pre-treatment on day 1) to day 13
  Part 2
CXCL10 in blood samples. | from Baseline (pre-treatment on day 1) to day 13
  Part 2

SECONDARY OUTCOMES:
Part 1-Safety, adverse events | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed on the number of reported adverse events
Part 1-Safety, laboratory values | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed on changes in laboratory values
Part 1-Safety, vital signs | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed on changes in vital signs
Part 1-Safety, lung function | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed on changes in lung function
Part 1-Safety, concomitant medication | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed on changes in concomitant medication
Part 1- Tolerability, adverse events | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed by reviewing adverse events
Part 1- Tolerability, laboratory values | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed by reviewing changes in laboratory values
Part 1- Tolerability, vital signs | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed by reviewing changes in vital signs
Part 1- Tolerability, lung function | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed by reviewing changes in lung function
Part 1- Tolerability, concomitant medication | from Baseline (pre-treatment on day 1) to day 7-10
  To be assessed by reviewing changes in concomitant medication
Part 1-Biomarker 1 | from Baseline (pre-treatment on day 1) to day 7-10
  Changes in sputum differential cell counts
Part 1-Biomarker 2 | from Baseline (pre-treatment on day 1) to day 7-10
  To evaluate and compare anti-viral IFN-stimulated genes in cells from expectorated sputum for SNG001 versus placebo
Part 2-Efficacy 1 changes in lung function | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare changes in lung function during the study period SNG001 with placebo
Part 2-Efficacy-2 BCSS score | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare BCSS score of SNG001 with placebo
Part 2-Efficacy-3 changes in BCSS symptom score | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare changes in BCSS symptom score during the study period of SNG001 with placebo
Part 2-Efficacy-4 return to normal (day to day) symptoms | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare time to return to normal (day to day) symptoms post a moderate exacerbation (Group B only) of SNG001 with placebo
Part 2-Efficacy-5 viral and bacterial load | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare sputum viral and bacterial load of SNG001 with placebo
Part 2-Efficacy-6 reliever medication usage | from Baseline (pre-treatment on day 1) to 13
  Evaluate and compare reliever medication usage during the treatment period of SNG001 with placebo
Part 2-Efficacy-7 antibiotic and oral corticosteroid usage | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare antibiotic and oral corticosteroid usage during the study period of SNG001 with placebo
Part 2-Efficacy-8 patient perceived efficacy | from Baseline (pre-treatment on day 1) to day 13
  Evaluate and compare patient perceived efficacy of SNG001 with placebo
Part 2-Safety, adverse event | from Baseline (pre-treatment on day 1) to day 28
  To be assessed on the number of reported adverse events
Part 2-Safety, laboratory values | from Baseline (pre-treatment on day 1) to day 28
  To be assessed on changes in laboratory values
Part 2-Safety, vital signs | from Baseline (pre-treatment on day 1) to day 28
  To be assessed on changes in vital signs
Part 2-Safety, concomitant medication | from Baseline (pre-treatment on day 1) to day 28
  To be assessed on changes in concomitant medication
Part 2- Tolerability, adverse events | from Baseline (pre-treatment on day 1) to day 28
  To be assessed by reviewing adverse events
Part 2- Tolerability, laboratory changes | from Baseline (pre-treatment on day 1) to day 28
  To be assessed by reviewing changes in laboratory values
Part 2- Tolerability, vital signs | from Baseline (pre-treatment on day 1) to day 28
  To be assessed by reviewing changes in vital signs
Part 2- Tolerability,concomitant medication | from Baseline (pre-treatment on day 1) to day 28
  To be assessed by reviewing changes in concomitant medication

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wilkinson, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (16):
- United Kingdom (16):
  - Celerion, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Tower Family Health Care, Bury
  - Lakeside Healthcare, Corby
  - Gartnavel General Hospital, Glasgow
  - Hemel Hempstead Hospital, Hemel Hempstead
  - Hull Royal Infirmary, Hull
  - Liverpool Heart and Chest Hospital, Liverpool
  - Queen Anne Medical Centre, London
  - Royal Brompton, London
  - Medicines Evaluation Unit, Manchester
  - North Tyneside General Hospital, North Shields
  - Nottingham University Hospital NHS Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - The Adam Practice, Upton

IPD SHARING:
Plan to Share IPD: Undecided